CLINICAL TRIAL: NCT02534558
Title: Pathomechanism of MicroRNA-29 in Shoulder Stiffness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IRB 102-5462B; ChangGungMH (Registry Identifier: ChangGungMH)
Record Dates: First submitted 2015-04-13; First posted 2015-08-27 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Stiffness of Shoulder, Not Elsewhere Classified
Keywords: MicroRNA-29; shoulder stiffness; mir-29a

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- miR-29a precursor oligonucleotide (Experimental): Effects of IL-1β, miR-29a precursor oligonucleotide treatment on the expressions of miR-29a, miR-29b or miR-29c in cell cultures are quantified
  Interventions: Biological: miR 29a
- miR-29a antisense oligonucleotide (Experimental): Effects of IL-1β, miR-29a antisense oligonucleotide treatment on the expressions of miR-29a, miR-29b or miR-29c in cell cultures are quantified
  Interventions: Biological: miR 29a

INTERVENTIONS:
Biological: miR 29a — Effects of IL-1β, miR-29a precursor or antisense oligonucleotide treatment on the expressions of miR-29a, miR-29b or miR-29c in cell cultures are quantified

SUMMARY:
The team integrates experimental analyses of clinical and basic medicine and transgenic mice models. miR-29a acts a potent protective factor against excessive fibrosis in myofibroblasts of subacromial bursa tissue. Gain of miR-29a stabilizes tendon and synovial tissue homeostasis that alleviates tissue stiffness and maintains function.

DETAILED DESCRIPTION:
Aims of first: The team will evaluate the associations among the mR-29a, miR-29b, miR-29c expression in subacromial bursa and subacromial fluid, incidence of shoulder stiffness, Constant scores, and VAS.

Aims of second: The team will isolate primary myofibroblast from subacromial bursa tissue as in vitro models and investigate the molecular events in the IL-1β modulation of miR-29a expression and the molecular mechanism underlying miR-29a inhibition of fibrotic matrix accumulation and apoptotic reactions in myofibroblast cultures.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 to 80 years
* receiving surgery for open acromioplasty

Exclusion Criteria:

* shoulder disorders caused by traumatic fracture
* previous surgery
* osteoarthritis
* malignant disorders
* hepatic disorders
* renal disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
The microRNA expression, mRNA expression as a measure | 48hr
  Differences among incidence, microRNA expression, mRNA expression of shoulder stiffness are analyzed using non-parametric student's t-test. P value of < 0.05 is considered statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Yang-Jih Ko, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No